CLINICAL TRIAL: NCT04008316
Title: Evaluation of Efficacy of Colchicine to Prevent Skin Relapses in Adult's IgA Vasculitis
Brief Title: Efficacy of Colchicine to Prevent Skin Relapses in Adult's IgA Vasculitis
Acronym: COLCHIVAS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P170910J; 2018-002114-13 (EudraCT Number)
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: IgA Vasculitis
MeSH Terms: conditions — IgA Vasculitis | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: prospective, controlled, double blind, randomized clinical trial: colchicine 1mg/day versus placebo for 6 months, with a 12 months total follow-up.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- colchicine 1mg/day (Experimental): Colchicine per os: 1 tablet (1mg) / day during 6 months
  Interventions: Drug: Colchicine
- placebo (Placebo Comparator): placebo 1 tablet / day during 6 months
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — colchicine 1mg/day

SUMMARY:
Immunoglobulin A vasculitis (IgA-V), formerly called Henoch-Schönlein purpura, is an immune vasculitis. Relapses are frequent (30%) and most of the time cutaneous (90%). Cutaneous involvement in adults is more severe (haemorrhagic blister or necrotic skin lesions) and more extensive than in children. Quality of life can be significantly altered by frequent cutaneous relapses. Colchicine, historically used for gout flares, is known to be an " old " low cost drug inducing very few adverse events. This molecule inhibits polymorphonuclear cell-chemotaxis to the site of inflammation explaining colchicine clinical efficacy in diseases such as Familial Mediterranean Fever or Behçet disease. Efficacy of colchicine has also been reported in cutaneous leukocytoclastic vasculitis including IgA-V, but without clinical studies supporting this attitude.

DETAILED DESCRIPTION:
Immunoglobulin A vasculitis (IgA-V), formerly called Henoch-Schönlein purpura, is an immune vasculitis. Relapses are frequent (30%) and most of the time cutaneous (90%). Cutaneous involvement in adults is more severe (haemorrhagic blister or necrotic skin lesions) and more extensive than in children. Quality of life can be significantly altered by frequent cutaneous relapses. Colchicine, historically used for gout flares, is known to be an " old " low cost drug inducing very few adverse events. It inhibits polymorphonuclear cell-chemotaxis to the site of inflammation explaining colchicine clinical efficacy in diseases such as Familial Mediterranean Fever or Behçet disease. Efficacy of colchicine has also been reported in cutaneous leukocytoclastic vasculitis including IgA-V, but without clinical studies supporting this attitude To assess efficacy of colchicine in adult's cutaneous IgA-V, the investigators conduct a prospective, controlled, double blind, randomized clinical trial, national, multicenter and multidisciplinary (internal medicine, nephrology and dermatology): colchicine 1mg/day versus placebo for 6 months, with a 12 months total follow-up. The primary objective is to evaluate efficacy of colchicine versus placebo to prevent cutaneous relapses, 6 months after inclusion, in adult patients with cutaneous IgA vasculitis alone or associated with non-severe digestive or renal involvement.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and < 85 years
2. IgA-V recently diagnosed (< 20 days since skin biopsy) and defined by :

   * Histologically proven small vessels vasculitis with IgA deposits IgA Vasculitis
   * Purpura and/or involvement of at least one organ among kidney, joint, or intestinal tract

Exclusion Criteria:

1. Severe renal IgA vasculitis:

   * impaired renal function, defined as an eGFR < 60 ml per minute per 1.73 m2 (MDRD or CKD-EPI formula)
   * proteinuria/creatinuria> 1g/g
   * Uncontrolled blood pressure (Systolic blood pressure > 170 mmHg, diastolic blood pressure > 100 mmHg)
2. Severe digestive IgA vasculitis:

   * intussusception
   * massive gastrointestinal haemorrhage (requiring transfusion)
   * intestinal ischemia
   * perforation
   * abdominal pain persisting more than one day (EVA > 5) and unresponsive to standard analgesics (level 1 or 2).
3. Prior (< 3 months) immunosuppressive or corticosteroid therapy
4. Additional cutaneous, and/or digestive and/or chronic renal diseases.
5. HIV and B and C Chronic hepatitis
6. Pregnancy or breast feeding or women without sufficient contraception among women of childbearing
7. Known allergy or intolerance to study medication or any of its excipients (lactose, saccharose)
8. Contraindication to colchicine such as:

   * severe hepatic insufficiency
   * combination with a macrolide (except spiramycin),
   * combination with pristinamycin
9. Participation in another interventional trial
10. Patient having not signed an informed consent
11. Patient without Social Security System Insurance

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2022-11-12 (Estimated); Study Completion 2023-05-12 (Estimated)

PRIMARY OUTCOMES:
the occurrence of the first cutaneous skin relapse | 6 months
  Cutaneous skin relapse is defined by reappearance of palpable purpura with lower limb predominance and not related to thrombocytopenia.

CONTACTS AND LOCATIONS:
Overall Officials: Evangeline PILLEBOUT, MD, Principal Investigator — APHP
Locations (1):
- Saint Louis Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided